CLINICAL TRIAL: NCT05176873
Title: A Phase 1 Study to Assess the Safety, Tolerability, Pharmacokinetics of DZD8586 in Healthy Adult Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dizal (Jiangsu) Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Dizal Pharmaceuticals (Industry)
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: DZ2021B0002
Record Dates: First submitted 2021-12-15; First posted 2022-01-04 (Actual); Last update posted 2023-09-07 (Actual); Status verified 2022-07

CONDITIONS: Lymphoma, Non-Hodgkin
MeSH Terms: conditions — Lymphoma, Non-Hodgkin

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Single dose of DZD8586 (Experimental): Single dose of DZD8586
  Interventions: Drug: DZD8586
- Single dose of Placebo (Placebo Comparator): Single dose of Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: DZD8586 — Single dose of DZD8586. Starting dose of DZD8586 is 20mg. If tolerated, subsequent cohorts will test increasing doses of DZD8586.
  Arms: Single dose of DZD8586
Drug: Placebo — A single oral dose of placebo will be given.
  Arms: Single dose of Placebo

SUMMARY:
This is a study in healthy adult participants. This is the first time this drug has ever been tested in human, and so it will help to understand what type of side effects may occur with this intervention. It will also measure the levels of drug in the body.

DETAILED DESCRIPTION:
This is a study in healthy adult participants. This is the first time this drug has ever been tested in human, and so it will help to understand what type of side effects may occur with this intervention. It will also measure the levels of drug in the body.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must be able to understand the nature of the trial and provide a signed and dated, written informed consent form before any study-specific procedures, sampling, and analyses.
2. Female and/or male aged 18~55 years (inclusive), at the time of signing the informed consent.
3. Body mass index (BMI) 18~30 kg/m2. Bodyweight of ≥ 45 kg (Female) or ≥ 55 kg (Male).
4. Non-smoker (never smoked or > 1 year from the last occurrence of smoking).
5. Participants are healthy as determined by medical history, physical examination, laboratory parameters, vital signs and ECG, performed before the first administration of the study drug, including the following criteria:

   * Normal AST, ALT, total bilirubin and serum alkaline phosphatase
   * Normal white blood cell (WBC), hemoglobin and platelet count
   * Normal coagulation function
   * CrCl ≥ 90 mL/min or eGFR > 80 mL/min/1.73m^2
   * QT/QTc interval < 450 ms
6. Male participants must be surgically sterile or using an acceptable method of contraception (defined as barrier methods in conjunction with spermicides) during the study (from the time they sign consent) and for 6 months after the last dose of the study drug to prevent pregnancy with a partner. Abstinence is an acceptable form of contraception, provided that the subject agrees to use barrier methods in conjunction with spermicides if they do engage in sexual intercourse.

   However, periodic abstinence, the rhythm method, and the withdrawal method are not acceptable methods of contraception. Male participants should refrain from sperm donation throughout this period.

   Female partners (of childbearing potential) of male participants must also use a highly effective method of contraception throughout this period.
7. Female participants must have negative pregnancy tests at screening and check-in AND: have been surgically sterile (with documentation of hysterectomy, bilateral oophorectomy, bilateral salpingectomy, bilateral tubal ligation/tubal occlusion) OR post-menopausal (no menstruation for a minimum of 12 months and confirmed by follicle-stimulating hormone (FSH) and serum estradiol at screening) OR, if of child-bearing potential, must be using an acceptable method of contraception such as an intrauterine device, implant or contraceptive injection, or two forms of the following (e.g. diaphragm, cervical cap, oral, patch or vaginal hormonal contraceptive, condom, spermicide, or sponge) for the last three months. All females must agree to continue to use their method of birth control for the duration of the study and a minimum of one complete menstrual cycle.

Exclusion Criteria:

1. Any condition which in the opinion of the investigator would interfere with the participant's ability to provide informed consent, comply with study instructions, confound interpretation of study results, or endanger the participant if he or she takes part in the trial.
2. Any of the following condition: positive Hepatitis B surface antigen (HBsAg), positive HCV antibodies, confirmed positive HIV test result, TB test or COVID-19 test.
3. History of malignancy of any type, except the following: surgically excised non-melanomatous skin cancers more than 5 years before receiving the study drug.
4. Has donated blood (including blood products) or experienced loss of blood ≥ 500 mL within 2 months before screening.
5. Reported history or any clinically significant abnormalities at the screening of cardiac, hepatic, renal, respiratory, GI, endocrine, immunological, dermatological, hematological, neurological, or psychiatrical disease.
6. Resting blood pressure > 140/90 mmHg at screening (a single repeat measurement is allowed if the initial measurement is outside of these limits). Resting pulse rate < 45 beats per minute.
7. Ingestion of grapefruit, grapefruit juice, pomegranate juice, star fruit, or orange marmalade (made with Seville oranges) within 1 week before screening.
8. Participation in another clinical study with an investigational product administered in the last 28 days.
9. Have previously completed or withdrawn from this study or any other study investigating DZD8586 and have previously received DZD8586.
10. Involvement in the planning and/or conduct of the study (applies to both Dizal staff and/or staff at the study site).
11. Previous enrolment or randomization in the present study.
12. For women only - currently pregnant (confirmed with positive pregnancy test) or breast-feeding.
13. Testing positive for alcohol and/or drugs of abuse at screening and check-in.
14. Self-reported substance abuse (e.g., alcohol, licit or illicit drugs) within 12 months of screening.
15. Unwilling or unable to limit the substance such as alcohol consumption as defined in the restriction section throughout the course of the study.
16. Received a live or live-attenuated vaccine within 3 months before the first dose of the study drug, except COVID-19 vaccine (within 2 weeks).
17. Use or intend to use any prescription within 28 days prior to study drug administration, unless deemed acceptable by the investigator (or designee). Concomitant prescription drugs should also be restricted during administration of study drug. Exceptions may be allowed on a case-by-case basis as agreed by the investigator and sponsor's medical monitor if considered not to interfere with the aims of the study.
18. Use or intend to use any nonprescription medications/products including vitamins, minerals, and phytotherapeutic/herbal/plant derived preparations, gastric pH modifiers, and neutralizing antacids within 14 days prior to study drug administration, unless deemed acceptable by the investigator (or designee). Concomitant non-prescription drugs should also be restricted during administration of study drug.
19. Use or intend to use slow-release medications/products considered to still be active within 14 days prior to check-in, unless deemed acceptable by the investigator (or designee).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2021-12-09 (Actual); Primary Completion 2022-05-11 (Actual); Study Completion 2022-05-22 (Actual)

PRIMARY OUTCOMES:
Number and percentage of participants with adverse event, serious adverse event, clinically defined abnormal vital signs, laboratory values, ECG abnormalities | 6 days after the last dose

SECONDARY OUTCOMES:
Plasma and urine concentrations of DZD8586 | 6 days after the last dose

CONTACTS AND LOCATIONS:
Overall Officials: Frank Lee, Principal Investigator — Frontage Clinical Services, Inc.
Locations (1):
- Frontage Clinical Service 200 Meadowlands Parkway, Secaucus, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No